CLINICAL TRIAL: NCT05093257
Title: Study of T Cells and Natural Killer Cells Expression in Patients With Immune Thrombocytopenic Purpura
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Mostafa Hashem, Resident of Clinical and Chemical Pathology, Sohag University
Other Study IDs: Soh-Med-21-10-12
Record Dates: First submitted 2021-10-12; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: T cells and NK cells in ITP patients
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: age and sex matched healthy control individuals.
  Interventions: Diagnostic Test: Laboratory investigations for control
- Group II: available number of ITP patients.
  Interventions: Diagnostic Test: Laboratory investigations for patients

INTERVENTIONS:
Diagnostic Test: Laboratory investigations for control — 1. Complete blood picture .
  2. Erythrocyte sedimentation rate(ESR).
  3. Liver function tests .
  4. Kidney function tests.
  5. CD3, CD4,CD8,CD16,CD56 from peripheral blood samples by Flowcytometry
  Groups: Group I
Diagnostic Test: Laboratory investigations for patients — 1. Complete blood picture .
  2. Erythrocyte sedimentation rate(ESR).
  3. Liver function tests .
  4. Kidney function tests.
  5. Anti-nuclear antibodies test by immunoflourescence for ITP patients.
  6. Bone marrow aspiration (for diagnosis of ITP).
  7. CD3, CD4,CD8,CD16,CD56 from peripheral blood samples by Flowcytometry.
  Groups: Group II

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune bleeding disorder characterized by bleeding due to isolated thrombocytopenia with platelet count less than 100 × 109/L. ITP is classified based on course of disease into acute (3- <12 months), and chronic (≥12 months). ITP usually has a chronic course in adults whereas approximately 80-90% of children undergo spontaneous remission within weeks to months of disease onset. The main pathogenesis of ITP is the loss of immune tolerance to platelet auto-antigens, which results in increased platelet destruction and impaired thrombopoiesis by autoantibodies and cytotoxic T lymphocytes (CTLs). Platelet autoantibodies, particularly antiglycoprotein (GP) GPIIbIIIa and anti-GPIbIX, are known to cause thrombocytopenia in patients with ITP. As a main component of cellular immunity, T cells play an important role in body defense and peripheral tolerance. Changing number and function of these cells is closely associated with various diseases, including ITP.NK cells can also modulate cellular immunity in ITP patients.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an autoimmune bleeding disorder characterized by bleeding due to isolated thrombocytopenia with platelet count less than 100 × 109/L.ITP is classified based on course of disease into acute (3- <12 months), and chronic (≥12 months). ITP usually has a chronic course in adults whereas approximately 80-90% of children undergo spontaneous remission within weeks to months of disease onset. The main pathogenesis of ITP is the loss of immune tolerance to platelet auto-antigens, which results in increased platelet destruction and impaired thrombopoiesis by autoantibodies and cytotoxic T lymphocytes (CTLs).Platelet autoantibodies, particularly antiglycoprotein (GP) GPIIbIIIa and anti-GPIbIX, are known to cause thrombocytopenia in patients with ITP. Auto-Abs production often occurs due to the loss of self-tolerance and increased stimulation of the immune system. The immune system includes a variety of B- and T cells which cooperate with each other in T-cell-dependent antibody production reactions and play significant roles in humoral and cellular immunity. Although the pathogenesis of ITP has not been clearly understood, the autoreactive B- and T cells have been directly and indirectly involved in Auto-Abs production, respectively. As a main component of cellular immunity, T cells play an important role in body defense and peripheral tolerance. Changing number and function of these cells is closely associated with various diseases, including ITP. It can be stated that CD4+ T cells are indirectly involved in ITP pathogenesis by inducing the increased activity of B cells during Auto-Abs production. Cytotoxic T lymphocytes (CTLs) are another subgroup of T lymphocytes characterized by the expression of CD8+ surface marker, destroying the pathogenic factors via granzyme and perforin production. These cells are increased in ITP patients and are involved in platelet destruction via augmented production of granzyme and perforin. NK cells can also modulate cellular immunity in ITP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with platelet less than 100 × 109/L diagnosed as immune thrombocytopenia according to bone marrow findings .

Exclusion Criteria:

* Other causes of thrombocytopenia as:

  * Hypersplenism.
  * Bone marrow diseases including : aplastic anemia, leukemia and myelodysplastic syndromes.
  * Cancer treatments like chemotherapy and radiation therapy.
  * Exposure to toxic chemicals as arsenic and benzene.
  * Medications to treat bacterial infections (antibiotics)and treat seizures or blood thinner heparin.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Group I: age and sex matched healthy control individuals. Group II: available number of ITP patients.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment the percentages of CD4+ cells from peripheral blood samples by Flowcytometry | within 3 days after collection of samples.
  Methods of the study: All patients were subjected to:
  1. Full history taking.
  2. Laboratory investigations:
     1. Complete blood picture .
     2. Erythrocyte sedimentation rate(ESR).
     3. Liver function tests .
     4. Kidney function tests.
     5. Anti-nuclear antibodies test by immunofluorescence for ITP patients.
     6. Bone marrow aspiration (for diagnosis of ITP).
     7. CD3, CD4 from peripheral blood samples by Flowcytometry.
Assessment the percentages of CD8+cells in ITP patients from peripheral blood samples by Flowcytometry . | within 3 days after collection of samples.
  Methods of the study: All patients were subjected to:
  1. Full history taking.
  2. Laboratory investigations:
     1. Complete blood picture .
     2. Erythrocyte sedimentation rate(ESR).
     3. Liver function tests .
     4. Kidney function tests.
     5. Anti-nuclear antibodies test by immunofluorescence for ITP patients.
     6. Bone marrow aspiration (for diagnosis of ITP).
     7. CD3, CD8 from peripheral blood samples by Flowcytometry.
Assessment the percentages of NK(CD16 +, CD56 +) cells in ITP patients from peripheral blood samples by Flowcytometry . | within 3 days after collection of samples.
  Methods of the study: All patients were subjected to:
  1. Full history taking.
  2. Laboratory investigations:
     1. Complete blood picture .
     2. Erythrocyte sedimentation rate(ESR).
     3. Liver function tests .
     4. Kidney function tests.
     5. Anti-nuclear antibodies test by immunofluorescence for ITP patients.
     6. Bone marrow aspiration (for diagnosis of ITP).
     7. CD16, CD56 from peripheral blood samples by Flowcytometry.